CLINICAL TRIAL: NCT01442363
Title: A Safety and Efficacy Study of BLI-1300 Ointment in Symptomatic Perianal Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment, discontinuation of program
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCD-02
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Perianal Crohn's Disease
Keywords: Crohn's disease; perianal; inflammatory bowel disease; fistula
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Fistula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BLI-1300 (low dose) (Experimental): Investigational Product (10%) Ointment
  Interventions: Drug: BLI-1300 low dose
- BLI-1300 (high dose) (Experimental): Investigational Product (20%) Ointment
  Interventions: Drug: BLI-1300 high dose
- placebo (Placebo Comparator): Placebo Ointment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: BLI-1300 low dose — topical ointment
  Arms: BLI-1300 (low dose)
Drug: BLI-1300 high dose — topical ointment
  Arms: BLI-1300 (high dose)
Drug: placebo — topical ointment
  Arms: placebo

SUMMARY:
This randomized, placebo-controlled, parallel, multi-center, double-blind pilot study is designed to determine the effects of BLI-1300 ointment on perianal pain associated with active Perianal Crohn's Disease (PCD).

ELIGIBILITY:
Inclusion Criteria:

* All subjects must give written informed consent.
* Male or female subjects, 18 years of age.
* Confirmed diagnosis of Crohn's Disease.
* Subject must have a 3 month documented history of perianal Crohn's Disease (PCD) and with clinical evidence of active PCD.
* Subject must have a Crohn's Disease Activity Index (CDAI) total score of ≤ 350 at Visit 2.
* Subjects must have a qualifying perianal pain score at Visits 1 and 2.

Exclusion Criteria:

* Women of childbearing potential who are not using adequate contraception.
* Women who are pregnant or breastfeeding.
* Subjects on unstable regimens of Crohn's therapy (e.g. tumor necrosis factor (TNF) inhibitors, immunosuppressants, steroids).
* Subjects taking strong analgesics that could interfere with pain measurements. Subjects with a perianal abscess requiring incision and drainage.
* Subjects with anal stenosis.
* Subjects with fistulae outside the immediate perianal area.
* Subjects who have had abdominal surgery for Crohn's disease within the past 12 weeks.
* Subjects who have had significant anorectal surgery for Crohns disease within the past 8 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, MPH, Study Director — Braintree Laboratories, Inc.
Locations (17):
- United States (17):
  - ACRI - Phase I, Anaheim, California
  - University of California - San Francisco, San Francisco, California
  - Borland Groover Clinic, Jacksonville, Florida
  - University of Maryland, Baltimore, Maryland
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - South Jersey Gastroenterology, Marlton, New Jersey
  - Long Island Clinical Research Associates, Great Neck, New York
  - New York Center for Clinical Research, Lake Success, New York
  - Mount Sinai Medical Center, New York, New York
  - Asheville Gastroenterology, Asheville, North Carolina
  - UNC School of Medical, Chapel Hill, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BLI-1300 (High Dose) | BLI-1300 (Low Dose) | Placebo
Started | 2 | 2 | 0
Completed | 2 | 1 | 0
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The study was discontinued and no patients were enrolled in the placebo arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | BLI-1300 (High Dose) | BLI-1300 (Low Dose) | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 0 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 0 | 4
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2
  Male | 1 | 1 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 2 | 0 | 4
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Perianal Pain Responders
Description: Percent of responders during Week 12. Response is defined as ≥30% decrease in mean NRS score for perianal pain (for the 7 treatment days immediately preceding the Week 12 visit) compared to the screening period.
Time Frame: 12 weeks
Population: The study was discontinued and no patients were enrolled in the placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | BLI-1300 (High Dose) | BLI-1300 (Low Dose) | Placebo
Number analyzed (Participants) | 2 | 2 | 0
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: The study was discontinued and no patients were enrolled in the placebo arm.
Arm/Group | BLI-1300 (High Dose) | BLI-1300 (Low Dose) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 1/2 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BLI-1300 (High Dose) (N=2) | BLI-1300 (Low Dose) (N=2) | Placebo (N=0)
rectal throbbing (Gastrointestinal disorders) | 0 | 1 | NA
diarrhea (Gastrointestinal disorders) | 0 | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sole disclosure restriction which sponsor imposes on the PI is a sixty (60) day limited restriction in order to the protect potentially proprietary information which may be patentable.